CLINICAL TRIAL: NCT03559296
Title: The Inter- and Intra-rater Reliability of Subcutaneous Echogenicity (SEG) Grade and Subcutaneous Echo-free Space (SEFS) Grade in Postmastectomy Lymphedema
Brief Title: Reliability of Subcutaneous Echogenicity (SEG) Grade and Subcutaneous Echo-free Space (SEFS) Grade
Status: Completed | Type: Observational
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Other Study IDs: 09.2018.466
Record Dates: First submitted 2018-06-06; First posted 2018-06-18 (Actual); Last update posted 2018-08-23 (Actual); Status verified 2018-08

CONDITIONS: Postmastectomy Lymphedema Syndrome
Keywords: imaging; assessment; edema; dermis; postmastectomy Lymphedema; reliability; ultrasound; grade
MeSH Terms: conditions — Edema; Breast Cancer Lymphedema

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study Group: patients with postmastectomy lymphedema who will undergo ultrasonographic assessment of postmastectomy lymphedema and circumferential tape measurement of arm
  Interventions: Diagnostic Test: Ultrasonographic assessment of postmastectomy lymphedema

INTERVENTIONS:
Diagnostic Test: Ultrasonographic assessment of postmastectomy lymphedema — Qualitative assessment of postmastectomy lymphedema via ultrasound (Subcutaneous echogenicity (SEG) and subcutaneous echo-free space (SEFS) grade systems for postmastectomy lymphedema) and circumferential tape measures ( The circumferential measurement of affected arm at MCP joint, wrist joint, 15 below elbow joint, elbow joint 15cm above elbow point) to assess upper extremity volume

SUMMARY:
The aims of this study is to determine the inter- and intra-rater reliability of SEG and SEFS grade systems for postmastectomy lymphedema.

DETAILED DESCRIPTION:
The clinical severity of lymphedema in an extremity is generally graded according to the International Society of Lymphology (ISL) stage. Stage 0 which refers to a latent or subclinical condition where swelling is not evident despite impaired lymph transport. It may exist months or years before overt edema occurs (Stages I-III). Stage I represents an early accumulation of fluid relatively high in protein content (e.g., in comparison with "venous" edema) and subsides with limb elevation. Pitting may occur. Stage II signifies that limb elevation alone rarely reduces tissue swelling and pitting is manifest. Late in Stage II, the limb may or may not pit as tissue fibrosis supervenes. Stage III encompasses lymphostatic elephantiasis where pitting is absent and trophic skin changes such as acanthosis, fat deposits, and warty overgrowths develop. Within each Stage, severity based on volume difference can be assessed as minimal (<20% increase) in limb volume, moderate (20-40% increase), or severe (>40% increase).

Because the ISL stage mainly consists of findings achieved by physical examinations and represents the most severely affected arm, it is subjective and may not reflect the distribution and mode of progression of the disease. The characteristic skin and subcutaneous tissue changes in extremities with chronic lymphedema are caused by changes in the extracellular matrix, such as connective tissue hypertrophy, fat accumulation resulting from both fat hypertrophy and an increased number of adipocytes, and interstitial protein-rich fluid accumulation. Ultrasound has been used to assess and diagnose lymphedema related changes. Subcutaneous echogenicity (SEG) and subcutaneous echo-free space (SEFS) grade systems for postmastectomy lymphedema are developed in order to grade lymphedema objectively and to delineate the disease status more clearly. However, the reliability of SEG and SEFS has not been evaluated. The aims of this study is to determine the inter- and intra-rater reliability of SEG and SEFS grade systems for postmastectomy lymphedema. Two physiatrist (one ten-year-experienced and one five-year-experienced in musculoskeletal ultrasonography) independently and alternately will assess the subjects once for each assessment. Three days later after the initial examination, one of the physiatrists reassessed the patients. The inter- and intra-rater reliability will be determined using kappa.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with unilateral postmastectomy lymphedema

Exclusion Criteria:

1. Bilateral lymphedema
2. The patients who had known systemic edemagenic conditions (e.g., cardiac/hepatic/renal failure, terminal cancer, on chemotherapy), and/or with cancer recurrence were excluded

Ages: 18 Years to 65 Years | Sex: Female
Age Groups: Adult, Older Adult
Gender Based: Yes — Women with postmastectomy lymphedema
Study Population: Women with postmastectomy lymphedema aged 18-65 years old
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2018-08-13 (Actual); Study Completion 2018-08-13 (Actual)

PRIMARY OUTCOMES:
International Society of Lymphology (ISL) stage by rater 1 | Day 0
  stage of the clinical severity of lymphedema
International Society of Lymphology (ISL) stage by rater 1 | Day 3
  stage of the clinical severity of lymphedema
International Society of Lymphology (ISL) stage by rater 2 | Day 0
  stage of the clinical severity of lymphedema

SECONDARY OUTCOMES:
MCP joint level affected arm | Day 0
  The circumferential measurement of affected arm at the metacarpophalangeal joints (MCP)
MCP joint level unaffected arm | Day 0
  The circumferential measurement of affected arm at the MCP joints
wrist joint level affected arm | Day 0
  The circumferential measurement of affected arm at wrist joint
wrist joint level unaffected arm | Day 0
  The circumferential measurement of affected arm at wrist joint
15 cm below the elbow joint point affected arm | Day 0
  The circumferential measurement of affected arm at 15 cm below the elbow joint point
15 cm below the elbow joint point unaffected arm | Day 0
  The circumferential measurement of affected arm at 15 cm below the elbow joint point
elbow joint point affected arm | Day 0
  The circumferential measurement of affected arm at the elbow joint point
elbow joint point unaffected arm | Day 0
  The circumferential measurement of unaffected arm at the elbow joint point
15 cm above the elbow joint point affected arm | Day 0
  The circumferential measurement of affected arm at 15 cm above the elbow joint point
15 cm above the elbow joint point unaffected arm | Day 0
  The circumferential measurement of affected arm at 15 cm above the elbow joint point
Affected extremity volume (mL) | Day 0
  Lymphedema of the limbs were assessed by a single physiotherapist using the circumferential and volumetric methods before and after the treatment protocol. The circumferential upper limb measurements were carried out with the arm abducted at 30°, starting at the level of the carpometacarpal joint, every 5 cm proximal to this point along both limbs. Then, a computer program (limb volumes professional version 5.0) was used to convert these values into limb volumes in milliliters.
Unaffected extremity volume (mL) | Day 0
  Lymphedema of the limbs were assessed by a single physiotherapist using the circumferential and volumetric methods before and after the treatment protocol. The circumferential upper limb measurements were carried out with the arm abducted at 30°, starting at the level of the carpometacarpal joint, every 5 cm proximal to this point along both limbs. Then, a computer program (limb volumes professional version 5.0) was used to convert these values into limb volumes in milliliters.
Subcutaneous echogenicity (SEG) grade by rater 1 | Day 0
  Grade 0: No increase in echogenicity in the subcutaneous layer. Namely, the subcutaneous fat layer is observed as black. Grade 1: Diffuse increase in echogenicity, but identifiable horizontal or obliquely oriented echogenic lines caused by connective tissue bundles. Grade 2: Diffuse increase in echogenicity. Echogenic lines are not identifiable
Subcutaneous echogenicity (SEG) grade by rater 1 | Day 3
  Grade 0: No increase in echogenicity in the subcutaneous layer. Namely, the subcutaneous fat layer is observed as black. Grade 1: Diffuse increase in echogenicity, but identifiable horizontal or obliquely oriented echogenic lines caused by connective tissue bundles. Grade 2: Diffuse increase in echogenicity. Echogenic lines are not identifiable
Subcutaneous echogenicity (SEG) grade by rater 2 | Day 0
  Grade 0: No increase in echogenicity in the subcutaneous layer. Namely, the subcutaneous fat layer is observed as black. Grade 1: Diffuse increase in echogenicity, but identifiable horizontal or obliquely oriented echogenic lines caused by connective tissue bundles. Grade 2: Diffuse increase in echogenicity. Echogenic lines are not identifiable
Subcutaneous echo-free space (SEFS) grade by rater 1 | Day 0
  Grade 0: No SEFS. Grade 1: Horizontally oriented (<45 degrees to the skin) SEFS only. Grade 2: Presence of vertically oriented (≥45 degrees to the skin) SEFS bridging the horizontally oriented SEFSs.
Subcutaneous echo-free space (SEFS) grade by rater 1 | Day 3
  Grade 0: No SEFS. Grade 1: Horizontally oriented (<45 degrees to the skin) SEFS only. Grade 2: Presence of vertically oriented (≥45 degrees to the skin) SEFS bridging the horizontally oriented SEFSs.
Subcutaneous echo-free space (SEFS) grade by rater 2 | Day 0
  Grade 0: No SEFS. Grade 1: Horizontally oriented (<45 degrees to the skin) SEFS only. Grade 2: Presence of vertically oriented (≥45 degrees to the skin) SEFS bridging the horizontally oriented SEFSs.

CONTACTS AND LOCATIONS:
Overall Officials: İlker Yagci, Prof, Msc, Principal Investigator — Marmara University; Esra Giray, MD, Principal Investigator — Marmara University
Locations (1):
- Marmara University School of Medicine Department of Physical Medicine and Rehabilitation, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
We don't plan to share.

REFERENCES:
- [Derived] Giray E, Yagci I. Interrater and Intrarater Reliability of Subcutaneous Echogenicity Grade and Subcutaneous Echo-Free Space Grade in Breast Cancer-Related Lymphedema. Lymphat Res Biol. 2019 Oct;17(5):518-524. doi: 10.1089/lrb.2018.0053. Epub 2018 Dec 20. PMID 30570358